CLINICAL TRIAL: NCT03090139
Title: Indicators of Sub-Optimal Response to Anti-Tumor Necrosis Factor (TNF) Therapy in Patients With Crohn's Disease (CD) and Ulcerative Colitis (UC): A Retrospective Chart Review in the Emerging Market (EM) Region (EXPLORE)
Brief Title: Sub-optimal Response to Anti-Tumor Necrosis Factor's in Inflammatory Bowel Disease in Emerging Markets
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: IBD-5001
Record Dates: First submitted 2017-03-22; First posted 2017-03-24 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Colitis, Ulcerative; Crohn Disease; Inflammatory Bowel Diseases
Keywords: Drug therapy
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Participants: All participants with diagnosis of UC and CD, who initiated treatment with anti-TNF therapy from 01 March 2010 up to 01 March 2015 will be observed. Retrospective data extraction will be done for eligible participants from March 2017 up to approximately February 2018.
  Interventions: Drug: Anti-TNF Therapy

INTERVENTIONS:
Drug: Anti-TNF Therapy — Anti-TNF therapy.

SUMMARY:
The purpose of this study is to establish the incidence of sub-optimal response to anti-TNF therapy in UC and CD participants.

DETAILED DESCRIPTION:
Participants with historical diagnosis of CD and UC who were naïve to anti-TNF therapy were observed in this retrospective study. The study will look to identify the local barriers in prescribing anti-TNF therapy, treatment patterns and indicators of sub-optimal response to anti-TNF therapy in UC and CD participants in real-world clinical practice in the EM countries, along with the associated incidence of sub-optimal response and impact on health care resource utilization (HCRU). The will enroll approximately 2000 participants.

The study consists of two periods, eligibility period followed by a data abstraction period. During the eligibility period participants who had initiated first anti-TNF therapy during 01 March 2010 up to 01 March 2015 will be recruited and observed. Participants will be followed up for a period of minimum 2 years (other than death) and a maximum of 5 years from the date of first treatment of anti-TNF therapy for CD and UC (Index date). During the data abstraction period participants who have eligible medical charts will be identified and all retrospective data will be collected.

This multi-center trial will be conducted in Argentina, China, Colombia, Mexico, Russia, Saudi Arabia, Singapore, South Korea, Taiwan and Turkey. The overall time to abstract data during the data extraction period from the web-based electronic data capture (EDC) system will be approximately 1 year from March 2017 to February 2018.

ELIGIBILITY:
Inclusion Criteria:

1. Who are 18 years or older at Index Date and diagnosed with UC or CD.
2. Who were naive to anti-TNF therapy and received their first dose of any anti-TNF therapy (index date) for UC or CD within the Eligibility Period from 01 March 2010 through 01 March 2015.

Exclusion Criteria:

1. Diagnosed with indeterminate/unspecified type of IBD.
2. Were part of an IBD-related clinical trial during the observational period should be excluded (that is, index date up to the date of chart abstraction).
3. Who received an anti-TNF therapy for any non-UC or non-CD conditions (example, rheumatoid arthritis, ankylosing spondylitis, psoriasis, or cancer).
4. Who received an anti-TNF/biologic therapy at any point that was administered outside of the labelled dosing regimen (example, episodic use of anti-TNF therapy).
5. With UC who had a total colectomy prior to their first anti-TNF therapy.
6. Charts not available.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of participants with a diagnosis of CD or UC who were naive to anti-TNF therapy and received their first dose of anti-TNF treatment for CD or UC during the eligibility period at private and public sites that routinely treat IBD participants and prescribe anti-TNF therapy from the targeted countries of interest.
Sampling Method: Non-Probability Sample
Enrollment: 1731 (Actual)
Dates: Start 2017-03-28 (Actual); Primary Completion 2018-06-13 (Actual); Study Completion 2018-06-13 (Actual)

PRIMARY OUTCOMES:
Incidence Rate of Sub-optimal Response in UC and CD Participants | 5 years
  Incidence rate will be calculated as the number of events divided by the total person time at risk, for participants under anti-TNF therapy.
Treatment Patterns in UC and CD Participants | 5 years
Number of Participants With Each Type of Anti-TNF Therapy | 5 years
Duration of Treatment | 5 years
Number of Participants With Response to Treatment | 5 years
  Number of participants with response to treatment will be assessed.
Treatment Pattern Results Stratified by Anti-TNF Response Group and by UC or CD Diagnosis | 5 years
  Treatment patterns results were as per the Anti-TNF therapy response from UC and CD participants.
Time-to-switch | 5 years
  The time to switch at which the participant switched to another anti-TNF therapy will be evaluated.
Time-to-first Indicator of Sub-optimal Therapy | 5 years
  Time-to-first indicator of sub-optimal therapy was defined as the occurrence of dose escalation, therapy augmentation, therapy switch, therapy discontinuation, hospitalization, or surgery of participant, which ever occurred first.

SECONDARY OUTCOMES:
Number of Participants With CD Achieving Clinical Response Based on Harvey Bradshaw Index (HBI) | Baseline up to 5 years
  Clinical response is defined as a decrease in HBI score of greater than or equal to (>=) 3 points from baseline. HBI score is used to measure the disease activity of CD. It consists of clinical parameters: abdominal pain (0-3, higher score means more severe pain), number of liquid stools per day, abdominal mass (0-3, where higher score means presence of swelling in the abdomen), and complications (score 1 per item). Total score is the sum of individual parameters. The score ranges from a minimum score of 0 to no pre-specified maximum score as it depends on the number of liquid stools, where higher scores indicating more severe disease.
Number of Participants With UC Achieving Clinical Response Based on Mayo Scores | Baseline up to 5 years
  Clinical response is defined as a decrease in the partial Mayo Score of at least 2 points and >=25% from baseline, with an accompanying decrease in rectal bleeding subscore of >=1 point from baseline or absolute rectal bleeding subscore of less than or equal to (<=) 1 point. Mayo score is an instrument designed to measure disease activity of UC. It consists of 3 subscores: stool frequency, rectal bleeding, and physician global assessment of disease severity, each graded from 0 to 3 with higher scores indicating more severe disease. These scores are summed to give a total score range of 0 to 9; where higher scores indicating more severe disease.
Number of Participants with Inflammatory Bowel Disease (IBD) Related Surgeries and Hospitalisation | 2 years prior to index anti-TNF therapy
  IBD-related surgeries and hospitalisation will be conducted in the two years prior to index anti-TNF therapy in UC or CD participants.
Number of Participants with Co-morbidities | Baseline
Number of Participants with Predictors of Sub-optimal Therapy in UC or CD Participants | Baseline up to 5 years
  The predictors of sub-optimal response will be assessed through multivariate analysis using logistic regression or other appropriate statistical methods. Multivariate analyses may be conducted to derive predictors of sub-optimal response to anti-TNF therapy globally and individually.
Health Care Resources Utilisation (HCRU) | Baseline up to 7 years
  HCRU will be calculated for physician clinic visits, emergency department visits, IBD-related surgeries, invasive procedures, imaging, and in-participant admissions related to UC or CD, or related complications as available in the medical record and captured in the electronic case report form (eCRF).
Physician Survey Questionnaire | Baseline
  The physician survey questionnaire will include questions on local accessibility to infusion centres, potential restrictions of prescription, potential local difficulties for drug access (example, reimbursement process, economic burden), and other reasons for participants compliant with the local label to not receive anti-TNF therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (76):
- Argentina (5):
  - Hospital Italiano, Ciudad Autonoma Buenos Aires, Buenos Aires
  - Hospital Italiano de La Plata, La Plata, Buenos Aires
  - Hospital Aleman, Ciudad Autonoma Buenos Aires
  - Hospital Britanico de Buenos Aires, Ciudad Autonoma Buenos Aires
  - Hospital Privado Centro Medico de Cordoba, Córdoba
- China (10):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - The Sixth Affiliated Hospital of Sun Yat-Sen University, Guangzhou, Guangdong
  - The Affiliated Drum Tower Hospital of Nanjing University, Nanjing, Jiangsu
  - First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Ruijin Hospital, Shanghai Jiaotong Uni. School of Med., Huangpu, Shanghai Municipality
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - No. 10 People's Hospital of Shanghai, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital affiliated with the Zhejiang University School of Medicine, Hangzhou, Zhejiang
- Colombia (5):
  - Hospital Militar Central, Bogotá
  - Hospital Universitario San Ignacio, Bogotá
  - Institucion Mediservis Tolima IPS S.A.S, Ibagué
  - Instituto de Coloproctologia ICO S.A.S., Medellín
  - Hospital Pablo Tobon Uribe, Medellín
- Mexico (6):
  - Investigacion Clinica de Leon S.C., León, Guanajuato
  - Centro de Investigacion Clinica Acelerada, S.C., Mexico City, Mexico City
  - Instituto Nacional de Ciencias Medicas y Nutricion Dr. Salvador Zubiran, Mexico City, Mexico City
  - Centro Regiomontano de Estudios Clinicos Roma S.C., Monterrey, Nuevo León
  - Centro de Investigacion y Manejo, Torre Medica Sanatorio Toluca, Toluca, State of Mexico
  - Hospital Medica Sur, Distrito Federal
- Russia (10):
  - The Saint Ioasaf Belgorod Regional Hospital, Belgorod
  - Irkutsk State Regional Hospital, Irkutsk
  - Kazan State Medical University, Kazan'
  - Moscow Clinical Research Center, Moscow
  - FSBI State Scientific Centre of Coloproctology" of the MoH of RF, Moscow
  - Moscow Region Research Cliniucal Institute, Moscow
  - Pokrovskaya Municipal Hospital, Saint Petersburg
  - Llc "Riat", Saint Petersburg
  - SBIH City Clinical Hospital #31, Saint Petersburg
  - FSBEI HE Stavropol State Medical University of Ministry of Healthcare of Russian Federation, Stavropol
- Saudi Arabia (6):
  - King Khalid National Guard Hospital, Jeddah
  - King Fahd General Hospital, Jeddah
  - King Fahd University Hospital, Khobar
  - King Khalid University Hospital, Riyadh
  - King Fahd Medical City, Riyadh
  - King Faisal Specialist Hospital & Research Center, Riyadh
- Singapore (5):
  - National University Cancer Institute,, Singapore
  - Singapore General Hospital- Parent, Singapore
  - CJ Ooi Gastroenterology Clinic Pte Ltd, Singapore
  - Tan Tock Seng Hospital, Singapore
  - Changi General Hospital- Parent, Singapore
- South Korea (10):
  - Yonsei University Wonju Severance Christian Hospital, Wŏnju, Gangwon-do
  - Hanyang University Guri Hospital, Guri-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon, Gyeonggi-do
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital, Yonsei University, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Taiwan (8):
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Chung Shan Medical University Hospital, Taichung
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan District
- Turkey (Türkiye) (11):
  - Ankara University Medical Faculty, Ankara
  - Turkiye Yuksek Ihtisas Training and Research Hospital, Ankara
  - Baskent University Ankara Hospital, Ankara
  - Gazi University Medical Faculty, Ankara
  - Gaziantep University Medical Faculty Sahinbey Educational Research Hospital, Gaziantep
  - Istanbul University Cerrahpasa Medical Faculty, Istanbul
  - Acibadem Fulya Hospital, Istanbul
  - Haydarpasa Numune Training and Research Hospital, Istanbul
  - Istanbul Medeniyet Uni Goztepe Training&Res Hosp, Istanbul
  - Izmir Katip Celebi Univ. Ataturk Training and Research Hospital, Izmir
  - Inonu Uni. Med. Fac., Malatya

REFERENCES:
- [Derived] Li J, Liu Z, Hu P, Wen Z, Cao Q, Zou X, Chen Y, Wang Y, Zhong J, Shen X, Demuth D, Fadeeva O, Xie L, Chen J, Qian J. Indicators of suboptimal response to anti-tumor necrosis factor therapy in patients from China with inflammatory bowel disease: results from the EXPLORE study. BMC Gastroenterol. 2022 Feb 4;22(1):44. doi: 10.1186/s12876-021-02074-z. PMID 35120446
- [Derived] Yamamoto-Furusho JK, Al Harbi O, Armuzzi A, Chan W, Ponce de Leon E, Qian J, Shapina M, Toruner M, Tu CH, Ye BD, Guennec M, Sison C, Demuth D, Fadeeva O, Khan QMR. Incidence of suboptimal response to tumor necrosis factor antagonist therapy in inflammatory bowel disease in newly industrialised countries: The EXPLORE study. Dig Liver Dis. 2020 Aug;52(8):869-877. doi: 10.1016/j.dld.2020.05.031. Epub 2020 Jun 17. PMID 32563721